CLINICAL TRIAL: NCT05996588
Title: Comparison Between Inhalational Anesthetic (Sevoflurane) and Intravenous Anesthetic (Propofol Infusion) for Maintenance of Sedation During Endoscopic Retrograde Cholangiopancreatography
Brief Title: Comparison Between Sevoflurane and Propofol for Maintenance of Sedation During ERCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Syed Muhammad Abbas, Associate Professor, Department of Anaesthesia, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIUT-ERC-2021/A-325
Record Dates: First submitted 2023-07-30; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Sedation Complication
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Propofol (Active Comparator): Propofol at a rate of 50 microgram/kg/min
  Interventions: Drug: Propofol 1 % Injectable Suspension
- Sevoflurane (Experimental): Sevoflurane inhalation with oxygen via nasal prongs at a concentration 4-5% to achieve a MAC of 0.25
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol 1 % Injectable Suspension — Propofol 1 % Injectable Suspension at a rate of 50 microgram/kg/min intravenously
  Other Names: Propofol
  Arms: Propofol
Drug: Sevoflurane — Sevoflurane inhalation anaesthetic at a concentration of 4-5% to achieve a MAC of 0.25
  Other Names: Sevoflurane inhalation anaesthetic
  Arms: Sevoflurane

SUMMARY:
After approval of ethical committee of Sindh Institute of Urology & Transplantation (SIUT), 86 patients were enrolled for the elective endoscopic retrograde cholangiopancreatography (ERCP). Randomization was done by a computer-generated randomization table. Patients were divided in two groups based on agents used for the research study. Both the groups were induced by injection midazolam 0.06 mg/kg body weight and injection nalbuphine 0.1 mg/kg body weight. In group A, anesthesia was maintained by Sevoflurane inhalation via nasal prongs with oxygen to achieve minimum alveolar concentration (MAC) approximately 0.25%. Whereas, in Group B propofol infusion at 50 ug/Kg/min started for maintenance of anaesthesia. Ketamine 0.5mg/kg intravenously was used to rescue the sedation level in both groups

DETAILED DESCRIPTION:
After approval of ethical committee of SIUT, 86 patients were enrolled for the elective endoscopic retrograde cholangiopancreatography (ERCP). Pre-operative assessment was done by history of patients, general physical examination, systematic examination, and laboratory investigations. Randomization was done by a computer-generated randomization table. Patients were divided in two groups based on agents used for the research study. Both the groups were induced by injection midazolam 0.06 mg/kg body weight and injection nalbuphine 0.1 mg/kg body weight. In group A, anesthesia was maintained by Sevoflurane inhalation via nasal prongs with oxygen to achieve minimum alveolar concentration (MAC) approximately 0.25%. Whereas, in Group B propofol infusion at 50 ug/Kilogram/min started for maintenance of anaesthesia.

When Ramsay Sedation Scale 5 is achieved then the endoscopist was allowed to insert endoscope. Injection Ketamine 0.5 mg/kg body weight was used for rescue sedation level. Upon arrival in operation theatre standard monitoring which includes pulse oximeter (SPO2), noninvasive blood pressure (NIBP), electrocardiogram (ECG) electrodes were applied, and baseline readings will be recorded. After that venous access was secured on a non-dominant hand by 20 Gauge IV cannula. Ringer's lactate or normal saline was then started at 8 ml/kg/hour and O2 was given by nasal prongs at 4 L/min. All baseline parameters were taken, after that readings were taken at 5 min, 10 min, 15 min, 20 min and so on till procedure ends.

Complications such as respiratory depression, coughing, gagging, nausea and vomiting were recorded during the procedure and treated accordingly. If SpO2 went down below 92% for more than 10 seconds or patient developed apnea, it was considered oxygen desaturation.

Oxygen desaturation was managed by O2 inhalation and supporting airway. A heart rate under 40 beats per minute was considered bradycardia and it will be managed by inj Atropine 10 ug/Kilogram intravenously (I/V). Mean arterial pressures level that is lower than 60 mmHg or 20% less than the baseline was regarded as hypotension and it was managed by fluid bolus or vasopressors.

After the procedure, patients were awakened and shifted to recovery room. Complications such as respiratory depression, coughing, gagging, nausea and vomiting were recorded and treated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age group of 20-60 years
* Both male and female patients.
* American Society of Anesthesiologist (ASA) physical status I-II
* Elective ERCP procedure.

Exclusion Criteria:

* Patients allergic to any study drug.
* American Society of Anesthesiology (ASA) Physical status III-IV
* Patients with uncontrolled Diabetes Mellitus,
* Hypertension and renal insufficiency.
* Body mass index (BMI) over 36 Kilogram/m2 (Morbid obesity)
* Obstructive Sleep Apnea
* Gastroesophageal reflux disease (GERD)
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Ramsay sedation score | 0-2 hours
  Clinical Score Patient's Characteristics
  1. Awake; agitated or restless or both
  2. Awake; cooperative, oriented, and tranquil
  3. Awake but responds to commands only
  4. Asleep; brisk response to light glabellar tap or loud auditory stimulus
  5. Asleep; sluggish response to light glabellar tap or loud auditory stimulus
  6. Asleep; no response to glabellar tap or loud auditory stimulus
Heart rate | 0-2 hours
  Heart rate via vitals monitoring device
Mean arterial blood pressure | 0-2 hours
  Mean arterial blood pressure via a non-invasive blood pressure monitor
Oxygen saturation | 0-2 hours
  Oxygen saturation via a pulse oximeter
Respiratory rate | 0-2 hours
  Respiratory rate via a vitals monitoring device

OTHER OUTCOMES:
Number of patients with post operative nausea | 0-2 hours
  Feeling of patient to vomit out
Number of patients with post operative vomiting | 0-2 hours
  Expulsion of stomach contents

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Q Abbas, FCPS, Study Chair — Professor Dept of Anaesthesiology
Locations (1):
- Syed Muhammad Abbas, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05996588/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05996588/SAP_001.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT05996588/ICF_002.pdf